CLINICAL TRIAL: NCT03046108
Title: Comparison Between Blind and Ultrasound Guided Injection in Morton Neuroma
Brief Title: Blind and Ultrasound Guided Injection in Morton Neuroma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complejo Hospitalario Universitario de Granada (Other)
Responsible Party: Principal Investigator, FERNANDO RUIZ SANTIAGO, PhD, section chief musculoskeletal radiology, Complejo Hospitalario Universitario de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0565-N-16
Record Dates: First submitted 2016-11-20; First posted 2017-02-08 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Morton Neuroma
MeSH Terms: conditions — Morton Neuroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- blind injection of Morton neuroma (Active Comparator): Percoutaneous blind injection in Morton neuroma by subcutaneous needle group 1 are going to be injected by an experimented orthopaedic surgeon based on anatomic landmark. There is no internal control of the needle placement.
  Mixture of 1 cc of 2% mepivacaine (Mepivacaina Normon 2%® )+ 40 mg of triamcinolone (Trigon Depot®) in each of the web spaces affected with Morton neuroma is injected.
  Up to 4 injections are allow in the first three months of follow-up
  Interventions: Device: blind injection of Morton neuroma; Drug: blind injection of Mepivacaine; Drug: blind injection of Triamcinolone
- blind injection of Mepivacaine (Active Comparator): 1 cc of 2% mepivacaine (Mepivacaina Normon 2%® )+ 40 mg of triamcinolone (Trigon Depot®) in each of the web spaces affected with Morton neuroma is injected.
  Up to 4 injections are allow in the first three months of follow-up
  Interventions: Device: blind injection of Morton neuroma; Drug: blind injection of Mepivacaine; Drug: blind injection of Triamcinolone
- blind injection of Triamcinolone (Active Comparator): 40 mg of triamcinolone (Trigon Depot®) in each of the web spaces affected with Morton neuroma is injected. Up to 4 injections are allow in the first three months of follow-up
  Interventions: Device: blind injection of Morton neuroma; Drug: blind injection of Mepivacaine; Drug: blind injection of Triamcinolone
- ultrasound guided injection (Experimental): US guided injection in Morton neuroma by subcutaneous needle. group 2 are going to be injected by an experimented musculoskeletal radiologist under ultrasound guidance. There is internal control of needle placement by ultrasound.
  Interventions: Device: ultrasound guided injection; Drug: guided injection of mepivacaine; Drug: guided injection of Triamcinolone
- guided injection of mepivacaine (Experimental): 2% mepivacaine (Mepivacaina Normon 2%® ) in each of the web spaces affected with Morton neuroma is injected.
  Up to 4 injections are allow in the first three months of follow-up
  Interventions: Device: ultrasound guided injection; Drug: guided injection of mepivacaine; Drug: guided injection of Triamcinolone
- guided injection of Triamcinolone (Experimental): 40 mg of triamcinolone (Trigon Depot®) in each of the web spaces affected with Morton neuroma is injected. Up to 4 injections are allow in the first three months of follow-up
  Interventions: Device: ultrasound guided injection; Drug: guided injection of mepivacaine; Drug: guided injection of Triamcinolone

INTERVENTIONS:
Device: blind injection of Morton neuroma — Introduction of a needle based in anatomical landmark
  Other Names: Blind introduction of the needle
  Arms: blind injection of Mepivacaine; blind injection of Morton neuroma; blind injection of Triamcinolone
Drug: blind injection of Mepivacaine — blind injection of 1 cc of Mepivacaine Normon 2% ®
  Arms: blind injection of Mepivacaine; blind injection of Morton neuroma; blind injection of Triamcinolone
Drug: blind injection of Triamcinolone — blind injection of 40 mg of triamcinolone (trigon depot ®)
  Other Names: Blind introduction of Triamcinolone
  Arms: blind injection of Mepivacaine; blind injection of Morton neuroma; blind injection of Triamcinolone
Device: ultrasound guided injection — Introduction of a needle based guided by ultrasound
  Other Names: guided introduction of the needle
  Arms: guided injection of Triamcinolone; guided injection of mepivacaine; ultrasound guided injection
Drug: guided injection of mepivacaine — ultrasound guided injection of 1 cc of Mepivacaine Normon 2% ®
  Other Names: guided perineural injection
  Arms: guided injection of Triamcinolone; guided injection of mepivacaine; ultrasound guided injection
Drug: guided injection of Triamcinolone — ultrasound guided injection of 40 mg of triamcinolone (trigon depot ®)
  Other Names: guided perineural injection
  Arms: guided injection of Triamcinolone; guided injection of mepivacaine; ultrasound guided injection

SUMMARY:
The aim of this work trial is to compare the effectiveness of blind and ultrasound guided injection for Morton neuroma in order to determine which is more appropriate as the initial procedure in conservative treatment

DETAILED DESCRIPTION:
This is a evaluator-blinded randomized trial. The final sample size has been calculated to be 100 patients. 50 of group 1 are going to be injected by an experimented orthopaedic surgeon based on anatomic landmark. 50 of group 2 are going to be injected by an experimented musculoskeletal radiologist under ultrasound guidance.

The inclusion criteria are clinical suspicion of Morton neuroma confirmed in ultrasound scan. Included patients are assessed clinically by VAS score, the Manchester Foot Pain and Disability Schedule (MFPDS), and a generic quality-of-life instrument, the EQ-5D.

Injection includes 1 cc of 2% mepivacaine and 40 mg of triamcinolone in each web space with Morton Neuroma. According evolution until 4 injections were allowed the first 2 months of follow-up, Follow up was performed by phone calls and/or scheduled consultations at 15 days, 1 month, 45 days, 2 months, 3 months, 6 months and 1 year.

Statistical analysis was performed by unpaired Student's t test

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of Morton neuroma confirmed in ultrasound scan
* Symptoms present more than six months
* The thickness of the nerve must be at least 2 mm in short axis and at least 5 mm in the longitudinal axis.

Exclusion Criteria:

* Contraindication for the use of corticosteroids or local anesthetics
* Presence of inflammatory arthropathy or neuropathy
* Skin lesions in the area
* diabetes mellitus
* Infiltration or previous surgery in the area
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS score) | 1 year
  Pain relieve

SECONDARY OUTCOMES:
Manchester foot pain and disability index | 1 year
  Disability measurement
Generic quality-of-life instrument, the EQ-5D | 1 year
  Quality of life measurement

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO RUIZ SANTIAGO, PhD, Study Director — COMPLEJO HOSPITALARIO UNIVERSITARIO GRANADA
Locations (1):
- Complejo Hospitalario Universitario Granada, Granada, SPA, Spain

IPD SHARING:
Plan to Share IPD: Yes
our idea is to publish the short term results and the long term results in order to influence management of this pathology. Tables and statistical analysis will be available for review and metaanalysis.

REFERENCES:
- [Result] Saygi B, Yildirim Y, Saygi EK, Kara H, Esemenli T. Morton neuroma: comparative results of two conservative methods. Foot Ankle Int. 2005 Jul;26(7):556-9. doi: 10.1177/107110070502600711. PMID 16045848
- [Result] Thomson CE, Beggs I, Martin DJ, McMillan D, Edwards RT, Russell D, Yeo ST, Russell IT, Gibson JN. Methylprednisolone injections for the treatment of Morton neuroma: a patient-blinded randomized trial. J Bone Joint Surg Am. 2013 May 1;95(9):790-8, S1. doi: 10.2106/JBJS.I.01780. PMID 23636185
- [Result] Mahadevan D, Attwal M, Bhatt R, Bhatia M. Corticosteroid injection for Morton's neuroma with or without ultrasound guidance: a randomised controlled trial. Bone Joint J. 2016 Apr;98-B(4):498-503. doi: 10.1302/0301-620X.98B4.36880. PMID 27037432
- [Result] Hassouna H, Singh D, Taylor H, Johnson S. Ultrasound guided steroid injection in the treatment of interdigital neuralgia. Acta Orthop Belg. 2007 Apr;73(2):224-9. PMID 17515235